CLINICAL TRIAL: NCT06819241
Title: Effectiveness of Self-Management of Blood Pressure on the Management of Resistant Hypertension
Brief Title: Self-Management of Blood Pressure in Resistant Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF24368A
Record Dates: First submitted 2025-01-13; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Resistant Hypertension
Keywords: resistant hypertension; self-management of blood pressure
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HBP self-management with AI chatbot support (Experimental): Self-monitoring of HBP combined with AI chatbot responses
  Interventions: Behavioral: AI chatbot support
- HBP self-management without AI chatbot support (Experimental): Self-monitoring HBP combined with telemonitoring and case management
  Interventions: Behavioral: telemonitoring and case management
- HBP-guided usual care (No Intervention)

INTERVENTIONS:
Behavioral: AI chatbot support — Integrating the practice of self-monitoring of HBP with the use of AI chatbot responses. This arm includes reminders for patients to monitor their BP and take antihypertensive medications, and involves tracking BP readings over time and offering feedback. Moreover, this arm offers physician-endorsed guidance on modifying the dosage of antihypertensive medication and implementing lifestyle adjustments. It offers education on hypertension and the potential side effects of medication, as well as assistance with medication refills and scheduling appointments.
  Arms: HBP self-management with AI chatbot support
Behavioral: telemonitoring and case management — Combining self-monitoring of HBP with telemonitoring and case management. This arm includes reminders for patients to monitor their BP and take antihypertensive medications, and involves tracking BP readings over time and offering feedback. Moreover, this arm offers physician-endorsed guidance on modifying the dosage of antihypertensive medication and implementing lifestyle adjustments. It offers education on hypertension and the potential side effects of medication, as well as assistance with medication refills and scheduling appointments.
  Arms: HBP self-management without AI chatbot support

SUMMARY:
The trial is a 12-month randomized, parallel-group study comparing three arms: (1) HBP self-management with AI chatbot support, (2) HBP self-management without AI chatbot support, and (3) usual care. The primary objective is to evaluate differences in blood pressure changes and medication compliance between groups at 6 and 12 months.

DETAILED DESCRIPTION:
Hypertension management Hypertension, characterized by persistently elevated BP, stands as a predominant risk factor for cardiovascular disease (CVD) and all-cause mortality worldwide. Its importance lies in its pervasive prevalence and significant contribution to the global burden of disease. Hypertension not only increases the risk of adverse cardiovascular events such as heart attack, stroke, and heart failure but also predisposes individuals to a spectrum of other health complications including chronic kidney disease, peripheral artery disease, and cognitive impairment. Furthermore, hypertension often coexists with various metabolic disorders such as diabetes mellitus and dyslipidemia, amplifying the overall cardiovascular risk. Addressing hypertension is thus imperative for public health initiatives aimed at reducing the burden of CVD and improving population health outcomes.

Hypertension represents a modifiable risk element. Effective management strategies for hypertension encompass lifestyle modifications, pharmacological interventions, and regular monitoring to achieve and maintain optimal BP levels. By recognizing the importance of hypertension and implementing comprehensive approaches to its prevention, diagnosis, and treatment, healthcare systems can mitigate its adverse effects and promote better cardiovascular health on a global scale.

Resistant hypertension Resistant hypertension represents a critical subset of hypertension that presents challenges in achieving adequate BP control despite treatment with multiple antihypertensive medications. Its importance lies in its association with heightened cardiovascular risk, including an increased likelihood of adverse events such as stroke, heart attack, and kidney disease. Effective management of resistant hypertension requires comprehensive evaluation, tailored treatment regimens, and close monitoring to mitigate these risks. Addressing resistant hypertension is crucial for optimizing patient outcomes and reducing the burden of cardiovascular morbidity and mortality.

Self-monitoring of BP Self-monitoring of BP holds paramount significance in the management of hypertension and related cardiovascular complications. This practice entails patients regularly measuring their BP outside of clinical settings, often using HBP monitoring devices. The importance of self-monitoring BP lies in its ability to provide healthcare professionals with a more comprehensive understanding of patients' BP patterns, facilitating personalized treatment plans tailored to individual needs. Additionally, self-monitoring empowers patients to actively engage in their healthcare by promoting awareness of their BP levels and fostering adherence to prescribed treatment regimens. Research indicates that incorporating self-monitoring into hypertension management strategies leads to more accurate diagnosis, optimized treatment adjustments, and improved BP control. Furthermore, self-monitoring enables early detection of fluctuations in BP, aiding in the prevention of hypertensive crises and associated complications such as stroke, heart attack, and kidney disease. Moreover, self-monitoring offers a cost-effective approach to hypertension management by reducing the need for frequent clinic visits and hospitalizations while enhancing patient satisfaction and autonomy. Overall, the integration of self-monitoring of BP into clinical practice represents a pivotal component of holistic hypertension care, offering numerous benefits in terms of patient outcomes, healthcare resource utilization, and long-term cardiovascular risk reduction. Therefore, the Taiwan Society of Cardiology and Taiwan Hypertension Society have embraced the 722 protocol as a standardized approach for HBP monitoring. The 722 protocol refers to duplicate BP readings taken per occasion ("2"), twice daily ("2"), over seven consecutive days ("7"). This protocol serves to validate hypertension diagnoses and to tailor antihypertensive medication adjustments accordingly.

Telemonitoring Telemonitoring plays a pivotal role in hypertension care by facilitating remote monitoring of patients' BP levels and treatment adherence. This approach enables healthcare providers to obtain real-time data on patients' BP readings, allowing for timely interventions and adjustments to treatment regimens as needed. By empowering patients to actively engage in self-management and promoting regular monitoring outside of clinical settings, telemonitoring helps to improve BP control and reduce the risk of cardiovascular complications associated with uncontrolled hypertension. Furthermore, telemonitoring enhances patient-provider communication and enables more personalized and proactive healthcare delivery, ultimately contributing to better patient outcomes in hypertension management.

Artificial intelligence chatbot The application of artificial intelligence (AI) chatbots in clinical settings represents a burgeoning area of research and implementation. These AI-driven conversational agents offer promising avenues for enhancing patient care through various functionalities, including symptom assessment, medication adherence support, and patient education. By leveraging natural language processing and machine learning algorithms, AI chatbots can interact with patients in real-time, providing personalized responses and recommendations. Moreover, AI chatbots have the potential to streamline administrative tasks, such as appointment scheduling and medical record retrieval, thereby improving workflow efficiency in healthcare settings. As the technology continues to evolve, the integration of AI chatbots holds immense potential for augmenting clinical decision-making processes and optimizing patient outcomes.

Investigational product(s)

1. HBP self-management with AI chatbot support: Integrating the practice of self-monitoring of HBP with the use of AI chatbot responses.
2. HBP self-management without AI chatbot support: Combining self-monitoring of HBP with telemonitoring and case management.

Both arms mentioned above include reminders for patients to monitor their BP and take antihypertensive medications. They also involve tracking BP readings over time and offering feedback. Moreover, these arms offer physician-endorsed guidance on modifying the dosage of antihypertensive medication and implementing lifestyle adjustments. They offer education on hypertension and the potential side effects of medication, as well as assistance with medication refills and scheduling appointments.

Risks

1. Technological barriers: Certain individuals, specifically elderly patients or those with limited proficiency in technology, may encounter difficulties when attempting to utilize the AI chatbot proficiently.
2. Privacy and data security: AI chatbots are utilized to gather and analyze sensitive health information. It is crucial to implement strong measures to guarantee the security and privacy of data.
3. Bias and inaccuracy: AI chatbots depend on algorithms that are trained using pre-existing data, which can potentially introduce bias or inaccuracies in the recommendations they offer. Regular surveillance and revisions of the chatbot's algorithms are imperative.

Benefits

1. Personalized support: Patients can be support from an AI chatbot or case manager by receiving personalized recommendations and reminders, potentially enhancing compliance to medication regimens and lifestyle changes.
2. Improved BP control: HBP self-management with and without AI chatbot support may lead to better BP control compared to usual care. This can reduce the risk of cardiovascular events such as heart attacks and strokes.
3. Reduced healthcare costs: Improved BP control and reduced healthcare utilization due to better self-management HBP may lead to cost savings for both patients and healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. receiving ≥3 antihypertensive medications of different classes, including a diuretic, and baseline BP >130/80 mmHg; or receiving ≥ 4 medications regardless of BP

Exclusion Criteria:

1. unable to conduct self-monitor BP because of cognitive dysfunction
2. poor adherence to medication
3. poor digital capabilities
4. pregnant
5. terminal disease
6. an acute cardiovascular event in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-02-16 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in HBP (systolic BP and diastolic BP) between baseline and each follow-up visit. | 6 and 12 months
  Primary endpoint

SECONDARY OUTCOMES:
Office blood pressure endpoint | 6 and 12 months
  Difference between intervention and control groups in change in office blood pressure (OBP; systolic BP and diastolic BP) between baseline and each follow-up visit.
Antihypertensive drug compliance endpoint | 6 and 12 months
  Difference between intervention and control groups in compliance to antihypertensive drugs during follow-up period, measured by pill count method.

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei